CLINICAL TRIAL: NCT01688245
Title: A Text Message Behavioral Intervention to Reduce Alcohol Consumption in Young Adults
Acronym: TRAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO12080344
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Alcohol Consumption; Alcohol Intoxication
Keywords: young adults; alcohol consumption; mobile health; text message
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): No SMS dialog
- SMS Assessments (Active Comparator): Weekly post-weekend drinking outcome assessments
  Interventions: Behavioral: SMS Assessments
- SMS Assessments & Feedback (Experimental): Weekly pre-weekend drinking intention & post-weekend drinking outcome assessments with personalized feedback and harm-reduction support
  Interventions: Behavioral: SMS Assessments & Feedback

INTERVENTIONS:
Behavioral: SMS Assessments & Feedback — Weekly pre-weekend drinking plan and post-weekend drinking outcome assessments with personlaized feedback
  Arms: SMS Assessments & Feedback
Behavioral: SMS Assessments — Weekly post-weekend drinking outcome assessments
  Arms: SMS Assessments

SUMMARY:
Investigators aim to test the effectiveness of a text-message-based behaivoral intervention in reducing binge drinking among young adults.

DETAILED DESCRIPTION:
Alcohol consumption, especially in the form of heavy episodic drinking (bingeing), is common among young adults. Despite high rates of illness and injury associated with heavy episodic drinking, many young adults are not aware of the risks, few seek help for their drinking and many at-risk are not exposed to prevention-based intervention. Opportunistic screening in hospital Emergency Departments (EDs) tied to behavioral interventions has the potential to prevent future alcohol-related harm among young adults, but efficacy across outcomes has been mixed and large-scale implementation of prevention programs is low. Given the rapidly growing use of cell phone text-messaging (SMS) as a primary form of communication among young adults, SMS could be used to deliver health prevention interventions. We will recruit young adults identified in the ED with hazardous drinking behavior in a 3-arm randomized controlled trial to test the hypothesis that exposure to a 12-week SMS program will result in immediate (3-month) and lasting (6-, and 9-month) decreases in alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* AUDIT-C score 3 or more for women and 4 or more for men

Exclusion Criteria:

* Current treatment for psychiatric disease
* Any prior treatment for drug or alcohol use disorder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 765 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Timeline Follow-back Procedure | 30 Days

SECONDARY OUTCOMES:
Injury Behavior Checklist | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Suffoletto, MD MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center-Mercy Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Suffoletto B, Kristan J, Chung T, Jeong K, Fabio A, Monti P, Clark DB. An Interactive Text Message Intervention to Reduce Binge Drinking in Young Adults: A Randomized Controlled Trial with 9-Month Outcomes. PLoS One. 2015 Nov 18;10(11):e0142877. doi: 10.1371/journal.pone.0142877. eCollection 2015. PMID 26580802
- [Derived] Suffoletto B, Callaway CW, Kristan J, Monti P, Clark DB. Mobile phone text message intervention to reduce binge drinking among young adults: study protocol for a randomized controlled trial. Trials. 2013 Apr 3;14:93. doi: 10.1186/1745-6215-14-93. PMID 23552023